CLINICAL TRIAL: NCT02275754
Title: Improving Quality of Life Among Hispanic/Latino Breast, Colorectal & Prostate Cancer Survivors: A Randomized Control Trial of Patient Navigators Using the LIVESTRONG Cancer Navigation Services Program
Brief Title: Redes III Patient Navigator Qol Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC20110094H; U54CA153511 (NIH)
Record Dates: First submitted 2014-09-15; First posted 2014-10-27 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PN+LCNC (Experimental): Patient Navigation plus LIVESTRONG Cancer Navigation Center (PN+LCNC): Participants assigned to this group will be assisted by the patient navigator with their health-related needs. The patient navigator will call the study participant on a weekly basis for the first three months of their participation in the study, and on a monthly basis thereafter to see if study participant needs anything pertaining to their cancer care.
  Interventions: Behavioral: PN+LCNC
- PN only (Active Comparator): Patient Navigation ONLY. Participants assigned to this group will be assisted by the patient navigator with their health-related needs. Navigation will occur ONLY on contact with navigators initiated by the study participants.
  Interventions: Behavioral: PN Only

INTERVENTIONS:
Behavioral: PN+LCNC — Patient Navigation plus LIVESTRONG Cancer Navigation Center (PN+LCNC): Participants assigned to this group will be assisted by the patient navigator with their health-related needs. The patient navigator will call the study participant on a weekly basis for the first three months of their participation in the study, and on a monthly basis thereafter to see if study participant needs anything pertaining to their cancer care.
  Arms: PN+LCNC
Behavioral: PN Only — Participants will be navigated by PN on request
  Arms: PN only

SUMMARY:
This proposed 5-year Redes En Acción research study involves a mixed-methods approach that occurs in two phases across two distinct and diverse HL communities. The RCT involves a 2 X 4 randomized repeated measures design with experimental condition (combined patient navigation [PN] over 3 months with access to LCNS PN services[PNLCNS] vs. a PN only condition) as the between-groups factor, and time-point (baseline/pre-randomization [T1]; post-PNLCNS [about 3-months post-T1; T2], and about 6- [T3] and about 12-months [T4] follow-up post-T2) as the within-groups factor; total follow-up is 15 months. The investigators will compare the effects of the PNLCNS and PN only conditions on QOL and treatment follow-up compliance in 300 (after attrition; n=100, Chicago and n=100, San Antonio) breast, colorectal and prostate HL cancer survivors with no evidence of metastatic disease.

DETAILED DESCRIPTION:
Hispanic/Latinos (HL) are the largest and fastest-growing minority population in the nation. HLs generally have lower survival rates for most cancers, even after accounting for differences in age and stage distribution, which may reflect less access to timely, high-quality treatment. They also experience disproportionately higher health disparities in quality of care and access to care. The experience of cancer survivorship is often characterized by significant challenges. Despite these challenges and significant disparities observed among HLs, there is very limited knowledge of survivorship-related issues and priorities among HLs, specifically the effectiveness of using promotores/patient navigators (PN) in linking HL cancer survivors with unmet psychosocial needs to appropriate psychosocial services. The existing community-based infrastructure of the Lance Armstrong Foundation (LAF) LIVESTRONG Cancer Navigation Services (LCNS) PN program provides an excellent opportunity to evaluate its efficacy in improving QOL among HLs. This proposed 5-year Redes En Acción research study involves a mixed-methods approach that occurs in two phases across two distinct and diverse HL communities. Phase I will use a community-based participatory research (CBPR) approach to engage community-based partners that provide services to breast, colorectal and prostate HL cancer survivors. In this phase, the investigators will gather community partners for action-oriented group meetings at each site to present components and targets of the combined PN and LCNS PN program (PNLCNS). Through this CBPR approach to generate valuable community feedback, the investigators will enhance the role of the PN, develop and extend existing cooperative relationships to facilitate participant recruitment, and prepare community-based partners to disseminate and implement the PNLCNS program upon the established efficacy of the proposed randomized controlled trial (RCT) of Phase II. Phase II will test a RCT to evaluate the efficacy of a culturally tailored PNLCNS program on improving general and disease-specific quality of life (QOL) and treatment follow-up compliance among breast, colorectal and prostate HL cancer survivors. Phase II also will evaluate the extent to which intervention-associated improvements in these outcomes are mediated by targets of the PNLCNS program (e.g., communication with medical team, meeting unmet needs and improving health behaviors). The RCT involves a 2 X 4 randomized repeated measures design with experimental condition (combined patient navigation [PN] over 3 months with access to LCNS PN services[PNLCNS] vs. a PN only condition) as the between-groups factor, and time-point (baseline/pre-randomization [T1]; post-PNLCNS [about 3-months post-T1; T2], and about 6- [T3] and about 12-months [T4] follow-up post-T2) as the within-groups factor; total follow-up is 15 months. The investigators will compare the effects of the PNLCNS and PN only conditions on QOL and treatment follow-up compliance in 300 (after attrition; n=100, Chicago and n=100, San Antonio) breast, colorectal and prostate HL cancer survivors with no evidence of metastatic disease. To understand the mechanisms by which the PNLCNS significantly impacts QOL and treatment compliance outcomes, the investigators also will examine changes in unmet cancer needs, communication with the medical team, health behaviors, psychological distress, worry, coping and general self-efficacy as potential mediators of the intervention effects. The investigators will also evaluate the extent to which other factors such as preparation for consultation (i.e., medical visit) and satisfaction with cancer care are associated with our QOL and treatment follow-up compliance outcomes. Study findings will fill a significant gap in our understanding of the extent to which PN programs and existing community-based resources targeting survivors can improve the QOL of a growing number of HL cancer survivors who experience an unequal burden of unmet needs after cancer treatment. The efficacy of the proposed RCT will provide a conceptually sound and clinically relevant approach to address the needs of HL cancer survivors by integrating evidence-based practice into existing community resources and infrastructure, thus facilitating the dissemination and translation of study findings through Phase I's CBPR process.

ELIGIBILITY:
Inclusion Criteria:

* Self identified Hispanic/Latino
* At least 18 yrs old
* Fluent in spoken Spanish or English
* Diagnosed with breast, prostate or colorectal cancer within the past fifteen months and thus considered a cancer survivor and are currently not undergoing treatment, with the exception of hormone therapy for prostate patients
* No evidence of metastatic disease
* No current severe mental illness
* No substance dependence within the past year -

Exclusion Criteria:

* Does not meet inclusion criteria
* Psychotic Disorder
* Active Suicidal Ideation
* Substance dependence (alcohol/drugs) within the past 12 months
* Does not meet the requisite cutoff of 3 or more correct responses on SPMSQ (Short Portable Mental Status Questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2015-09 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
General quality of life | 15 months
  The Functional Assessment of Cancer Therapy-General (FACT-G) will be administered to evaluate general domains of QOL. The FACT-G, now in its fourth revision, is one of the most widely used instruments to assess overall adjustment to cancer treatment and survivorship. It is a 27-item self-report questionnaire that takes less than 15 minutes to administer. The FACT-G assesses QOL in four domains of well-being: physical, social/family, emotional and functional well-being. Patients are asked to indicate the extent to which they agree with statements such as "I have pain," "I feel ill," "I get emotional support from my family," "I get support from my friends," "I feel sad," "I feel nervous," "I am sleeping well," and "I am content with the quality of my life right now." The scale is validated for use in many settings with many age groups. We will calculate a composite score for general QOL as well as subscale scores for specific domains of QOL.
Disease specific quality of life | 15 months
  We will administer three cancer-specific FACT versions, the FACT-B (breast cancer survivors), FACT-C (colorectal cancer survivors) or FACT-P (prostate cancer survivors). Each version addresses QOL issues that are common sequelae of that certain cancer. For example, the FACT-P evaluates concerns on sexuality, pain, and bowel and bladder function, the FACT-C asks questions about bowel movement control, weight loss and cramping in the abdominal area, and the FACT-B inquires about hair loss, shortness of breath and swelling in the arms. Reliability of the FACT-G, as well as all cancer site-specific FACT measures are acceptable (Cronbach's α>.70). Composite scores for disease-specific QOL will be calculated across each cancer site. Cancer site specific modules scores are standardized and can be combined across cancer sites.
Treatment Follow-up compliance | 15 months
  Because all of our HL cancer survivors will be recruited within 12-months post-treatment completion for a primary tumor, we will follow ACS guidelines for follow-up care for one- to two-years post-treatment. We will assess via self-report whether the participant missed a scheduled follow-up appointment during the study period. A compliance categorical outcome measure (compliant vs. non-compliant) will be calculated for each participant. Compliance will be defined as attending all scheduled follow-up appointments specific to cancer treatment follow-up during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie G Ramirez, DrPH, Principal Investigator — The University of Texas Health Science Center at San Antonio; Frank Penedo, PhD, Study Director — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Noriega Esquives BS, Moreno PI, Munoz E, Lad TE, Hollowell CMP, Benzo RM, Ramirez AG, Penedo FJ. Effects of a culturally tailored patient navigation program on unmet supportive care needs in Hispanic/Latino cancer survivors: A randomized controlled trial. Cancer. 2025 Jan 1;131(1):e35626. doi: 10.1002/cncr.35626. Epub 2024 Nov 1. PMID 39487386